CLINICAL TRIAL: NCT06653972
Title: Efficacy and Safety of Liposomal Doxorubicin Combined with Vinorelbine in the Treatment of Advanced Metastatic Breast Cancer: a Single-Center, Prospective Phase II Clinical Study
Brief Title: Efficacy and Safety of a Two-week Dosing Regimen of Vinorelbine Combined with Liposomal Doxorubicin in the Treatment of HER2-negative Advanced Breast Cancer
Acronym: EASOVCWDITHABC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wang Jiayu (Other)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Wang Jiayu, doctor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC-015985
Record Dates: First submitted 2024-09-25; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-09

CONDITIONS: Her2-negative Metastatic Breast Cancer; Vinorelbine; Liposomal Doxorubicin
MeSH Terms: interventions — liposomal doxorubicin; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PLD+NVB (Experimental): Pegylated Liposomal Doxorubicin 25mg/m2 ivgtt d1 + vinorelbine25mg/m2 ivgtt d1/q14d.
  Interventions: Drug: Pegylated Liposomal Doxorubicin + vinorelbine,every cycle is 14d.

INTERVENTIONS:
Drug: Pegylated Liposomal Doxorubicin + vinorelbine,every cycle is 14d. — Pegylated Liposomal Doxorubicin 25mg/m2 ivgtt d1 + vinorelbine25mg/m2 ivgtt d1/q14d.

SUMMARY:
With advancements in various treatment modalities, the survival of breast cancer patients has continuously improved. Patients with advanced breast cancer who have undergone multiple lines of therapy still have treatment options, but standard treatment protocols are lacking. Anthracyclines are a cornerstone in breast cancer treatment; however, their cumulative dose-related cardiac toxicity limits their use. Liposomal doxorubicin exhibits comparable efficacy to conventional anthracyclines and is not affected by previous cumulative doses. The combination of vinorelbine with liposomal doxorubicin shows reduced cross-toxicity, and several studies have demonstrated the effectiveness of this regimen in metastatic HER2-negative breast cancer patients.

Therefore, we aim to explore whether optimizing the dosage and treatment cycle of this combination therapy can provide a viable treatment option for metastatic HER2-negative breast cancer patients who have previously received second-line or higher chemotherapy, seeking a regimen that balances efficacy and safety.

This study is a single-center, single-arm Phase II clinical trial planned to enroll 30 metastatic HER2-negative breast cancer patients who have previously undergone second-line or higher chemotherapy. Participants will receive an optimized regimen of liposomal doxorubicin combined with vinorelbine, with safety assessed every cycle and efficacy evaluated every three cycles. Treatment will continue until radiographic evidence indicates disease progression, intolerable toxicity occurs, informed consent is withdrawn, or the investigator decides to discontinue treatment. Following treatment, each participant will undergo survival follow-up every three months until death, loss to follow-up, or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old，and ≤70 years old.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
3. Expected survival period not less than 12 weeks.
4. At least 1 measurable lesion according to RECIST 1.1 standard.
5. Previously received treatment with taxanes and anthracyclines. Note: Taxanes and anthracyclines can be utilized at various treatment stages, including neoadjuvant/adjuvant，recurrence/metastasis, with a treatment duration of at least 2 cycles (e.g., 21 days/cycle). If disease progression or intolerance occurs during a treatment regimen containing taxanes or anthracyclines, prior usage does not need to meet the above criteria.
6. Patients with metastatic breast cancer have received ≥2 lines of chemotherapy. Note: The number of chemotherapy lines refers to chemotherapy agents(each regimen counting as one line, excluding endocrine therapies; maintenance therapy does not count toward the line number).

6. Immunohistochemistry (IHC) and fluorescence in situ hybridization (FISH) validated HER2 negative, including IHC- and IHC 1+/2+ with FISH negative.

7. The organ function must meet the following requirements：

1. . Blood Routine

   * ANC≥1.5×109/L；
   * PLT≥90×109/L；
   * Hb≥90 g/L；
2. . Blood Biochemistry

   * TBIL≤1.5×ULN；
   * ALT and AST≤2×ULN；ALT和AST≤5×ULN for patients with liver metastasis；
   * BUN and Cr≤1.5×ULN and the Creatinine Clearance Rate ≥50 mL/min (Cockcroft-Gault formula calculated)；
3. . Echocardiogram

   • LVEF≥50%；
4. . electrocardiogram

   * The QT interval (QTcF) corrected by Fridericia method less than 450 ms for male and less than 470 ms for female.

     8. Volunteer to join this study, sign informed consent, have good compliance and be willing to cooperate with follow-up.

Exclusion Criteria:

1. There is a third interstitial fluid accumulation that cannot be controlled by drainage or other methods (such as a large amount of hydrothorax and ascites).
2. Symptomatic or uncontrolled brain or meningeal metastases.
3. Patients with only bone or skin metastasis as the assessable lesion.
4. Previously suffered from other malignant tumors.
5. Those who have used vinorelbine or Pegylated Liposomal Doxorubicin during the advanced disease stage.
6. Individuals with a known history of allergies to the components of the interventions; History of immunodeficiency, including HIV positive, other acquired or congenital immunodeficiency diseases and a history of organ transplantation.
7. Any heart disease or other conditions evaluated unsuitable by the researcher.
8. Pregnant and lactating female patients, female patients with fertility and positive baseline pregnancy test results, or female patients of reproductive age who are unwilling to take effective contraceptive measures throughout the trial period.
9. According to the investigator's judgment, there are concomitant diseases that seriously endanger the patient's safety or affect the patient's completion of the study (including severe bleeding tendency, history of surgery within 2 weeks, hypertension beyond drug control, serious diabetes, active infection, thyroid disease, etc.).
10. Having a clear history of neurological or mental disorders, including epilepsy or dementia.
11. According to the RECIST 1.1 criteria, researchers determined that patients who received the last anti-tumor regimen before enrollment did not experience disease progression.
12. Immunohistochemistry (IHC) and fluorescence in situ hybridization (FISH) validated human epidermal growth factor receptor 2 (HER2) positive.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | Radiological examinations will be conducted every three cycles: at the end of Cycle 3, 6, 9,...(each cycle is 14 days). The PFS will last until disease progression，up to 2 years.
  PFS is defined as the time from randomization to the date of confirmed radiological progression or death from any cause.

SECONDARY OUTCOMES:
overall survival (OS) | The long-time survival will be followed every 3 months after the end of treatment,up to 5 years.
  OS is defined as the time from randomization to the date of death from any cause and censored at the date of final contact for patients who were still alive.
objective response rate (ORR) | Time Frame: Radiological examinations will be conducted every three cycles: at the end of Cycle 3, 6, 9, ......(each cycle is 14 days),assessed until cycle 15 . The efficacy will be evaluated according to RECIST 1.1 standard.
  ORR is defined as the proportion of patients with best response of complete response (CR) and partial response (PR) according to RECIST 1.1 standard.
clinical benefit rate (CBR) | Radiological examinations will be conducted every three cycles,at the end of cycle 3,6,9... (each cycle is 14 days).The efficacy will be evaluated according to RECIST 1.1 standard.
  CBR is defined as the proportion of patients with best response of complete response (CR) , partial response (PR) and stable disease (SD) according to RECIST 1.1 standard.
Disease Control Rate（DCR） | Radiological examinations will be conducted every three cycles,at the end of cycle 3,6,9... (each cycle is 14 days).The efficacy will be evaluated according to RECIST 1.1 standard.
  It is defined as the proportion of patients who achieve either a complete response (CR), a partial response (PR), or stable disease (SD) after treatment.
Time to Progression（TTP） | Radiological examinations will be conducted every three cycles: at the end of Cycle 3, 6, 9......(each cycle is 14 days). The TTP will last until disease progression,up to 2 years.
  It is the duration from the start of treatment until the disease shows signs of progression, such as tumor growth or the emergence of new lesions.

OTHER OUTCOMES:
treatment-related adverse events (TRAE) | Adverse events will be assessed every cycle (each cycle is 14 days) and graded according to the Common Terminology Criteria Adverse Events (CTCAE) version 5 until 1 month after the end of treatment.
  TRAE is defined as the adverse reactions that occur during the use of medication for treatment and are supposed to be related to the intervention drugs.
quality of life (QoL) | The life quality questionnaire is arranged at baseline and every 3 months after enrollment until 6 months after the end of treatment.
  QoL assessment is examined by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire core 30 (EORTC QLQ-C30), of which 30 items were included. Items 1-28 are divided into 4 levels, with ratings ranging from 1 to 4 (the higher score indicates worse life quality). Items 29 and 30 are divided into 7 levels, with ratings ranging from 1 to 7 (the higher score indicates better life quality).

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: After the final analysis of this study on October 2026